CLINICAL TRIAL: NCT03515005
Title: Using Lay Health Advisors to Help African Americans Address the Social Context of Hypertension Management
Brief Title: Using Lay Health Advisors to Improve Hypertension Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment target not reached
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Daryl Thornton, MD, Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB18-00038
Record Dates: First submitted 2018-03-29; First posted 2018-05-03 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
Keywords: Hypertension; Community Health Workers; Community-Based Participatory Research; Health Equity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lay Health Advisors (Experimental): Intervention patients will meet monthly in small groups with a trained Lay Health Advisor.
  Interventions: Behavioral: Lay Health Advisor
- Usual Care (No Intervention): Control patients will receive usual care from their doctors.

INTERVENTIONS:
Behavioral: Lay Health Advisor — Patients will meet regularly Lay Health Advisors who will address the social context of their hypertension.
  Arms: Lay Health Advisors

SUMMARY:
Hypertension disproportionately affects and is inadequately controlled among African American and poor populations. The investigators propose to determine the impact of using trained lay health advisors to help patients address social contextual factors that influence the management of hypertension.

DETAILED DESCRIPTION:
Hypertension disproportionately affects and is inadequately controlled among African American and poor populations. Health providers generally lack the skills and resources to address social contextual factors (i.e. health and community services, social networks, social stressors, physical environment, and economic resources) that influence management of hypertension. Instead, providers tend to focus on adjusting antihypertensive medication prescriptions and exhorting patients to exercise and eat better. The investigators propose to determine the impact of using trained lay health advisors to help patients address social contextual factors that influence the management of hypertension. Helping patients address these barriers may lead not only to improved blood pressure but also to increased survival, reduced organ damage, and decreased health care costs. This project may also serve as a model of healthcare delivery innovation that could be used to address other health disparity conditions.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 outpatient blood pressures with systolic >140 or diastolic >90 mm Hg in last 6 months. Separate occurrences at least 1 day apart
* Age 18-59 years
* Non-diabetic
* Preserved kidney function (glomerular filtration rate >60 ml/min)
* English speaking

Exclusion Criteria:

* Mentally incompetent
* Pregnant
* Terminal illness
* Active substance abuse
* Documented coronary, peripheral arterial, or cerebrovascular disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | 1 year
  Difference between final and initial systolic and diastolic blood pressure readings

SECONDARY OUTCOMES:
Change in quality of life. | 1 year
  Differences in quality of life between final and initial measurements using the 12 item short form survey (SF-12). The SF-12 provides physical and mental health composite scores ranging from 0 (lowest level of health) to 100 (highest level of health)

CONTACTS AND LOCATIONS:
Overall Officials: John D Thornton, MD, MPH, Principal Investigator — MetroHealth System, Ohio
Locations (1):
- The MetroHealth System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egan BM, Li J, Hutchison FN, Ferdinand KC. Hypertension in the United States, 1999 to 2012: progress toward Healthy People 2020 goals. Circulation. 2014 Nov 4;130(19):1692-9. doi: 10.1161/CIRCULATIONAHA.114.010676. Epub 2014 Oct 20. PMID 25332288
- [Background] James SA, Van Hoewyk J, Belli RF, Strogatz DS, Williams DR, Raghunathan TE. Life-course socioeconomic position and hypertension in African American men: the Pitt County Study. Am J Public Health. 2006 May;96(5):812-7. doi: 10.2105/AJPH.2005.076158. Epub 2006 Mar 29. PMID 16571689
- [Background] Matthews KA, Kiefe CI, Lewis CE, Liu K, Sidney S, Yunis C; Coronary Artery Risk Development in Young Adults Study (CARDIA). Socioeconomic trajectories and incident hypertension in a biracial cohort of young adults. Hypertension. 2002 Mar 1;39(3):772-6. doi: 10.1161/hy0302.105682. PMID 11897761
- [Background] Cook S, Drum ML, Kirchhoff AC, Jin L, Levie J, Harrison JF, Lippold SA, Schaefer CT, Chin MH. Providers' assessment of barriers to effective management of hypertension and hyperlipidemia in community health centers. J Health Care Poor Underserved. 2006 Feb;17(1):70-85. doi: 10.1353/hpu.2006.0021. PMID 16520513
- [Background] Mercuri M, Sherbino J, Sedran RJ, Frank JR, Gafni A, Norman G. When guidelines don't guide: the effect of patient context on management decisions based on clinical practice guidelines. Acad Med. 2015 Feb;90(2):191-6. doi: 10.1097/ACM.0000000000000542. PMID 25354075
- [Background] Borzecki AM, Oliveria SA, Berlowitz DR. Barriers to hypertension control. Am Heart J. 2005 May;149(5):785-94. doi: 10.1016/j.ahj.2005.01.047. No abstract available. PMID 15894958
- [Background] Hill MN, Bone LR, Hilton SC, Roary MC, Kelen GD, Levine DM. A clinical trial to improve high blood pressure care in young urban black men: recruitment, follow-up, and outcomes. Am J Hypertens. 1999 Jun;12(6):548-54. doi: 10.1016/s0895-7061(99)00007-2. PMID 10371363
- [Background] Dennison CR, Post WS, Kim MT, Bone LR, Cohen D, Blumenthal RS, Rame JE, Roary MC, Levine DM, Hill MN. Underserved urban african american men: hypertension trial outcomes and mortality during 5 years. Am J Hypertens. 2007 Feb;20(2):164-71. doi: 10.1016/j.amjhyper.2006.08.003. PMID 17261462
- [Background] Rose LE, Kim MT, Dennison CR, Hill MN. The contexts of adherence for African Americans with high blood pressure. J Adv Nurs. 2000 Sep;32(3):587-94. doi: 10.1046/j.1365-2648.2000.01538.x. PMID 11012800
- [Background] Russell E, Johnson B, Larsen H, Novilla ML, van Olmen J, Swanson RC. Health systems in context: a systematic review of the integration of the social determinants of health within health systems frameworks. Rev Panam Salud Publica. 2013 Dec;34(6):461-7. PMID 24569976
- [Background] Wong K, Smalarz A, Wu N, Boulanger L, Wogen J. The association between hypertension-specific care management processes and blood pressure outcomes in US-based physician organizations. J Am Soc Hypertens. 2011 Nov-Dec;5(6):505-12. doi: 10.1016/j.jash.2011.08.002. Epub 2011 Oct 1. PMID 21958468
- [Background] Jackson EJ, Parks CP. Recruitment and training issues from selected lay health advisor programs among African Americans: a 20-year perspective. Health Educ Behav. 1997 Aug;24(4):418-31. doi: 10.1177/109019819702400403. PMID 9247822
- [Background] Dye CJ, Williams JE, Evatt JH. Improving hypertension self-management with community health coaches. Health Promot Pract. 2015 Mar;16(2):271-81. doi: 10.1177/1524839914533797. Epub 2014 May 16. PMID 24837989
- [Background] Margolius D, Bodenheimer T, Bennett H, Wong J, Ngo V, Padilla G, Thom DH. Health coaching to improve hypertension treatment in a low-income, minority population. Ann Fam Med. 2012 May-Jun;10(3):199-205. doi: 10.1370/afm.1369. PMID 22585883
- [Background] Brownstein JN, Chowdhury FM, Norris SL, Horsley T, Jack L Jr, Zhang X, Satterfield D. Effectiveness of community health workers in the care of people with hypertension. Am J Prev Med. 2007 May;32(5):435-47. doi: 10.1016/j.amepre.2007.01.011. PMID 17478270
- [Background] Krieger J, Collier C, Song L, Martin D. Linking community-based blood pressure measurement to clinical care: a randomized controlled trial of outreach and tracking by community health workers. Am J Public Health. 1999 Jun;89(6):856-61. doi: 10.2105/ajph.89.6.856. PMID 10358675
- [Background] Connell P, Wolfe C, McKevitt C. Preventing stroke: a narrative review of community interventions for improving hypertension control in black adults. Health Soc Care Community. 2008 Mar;16(2):165-87. doi: 10.1111/j.1365-2524.2007.00737.x. PMID 18290982
- [Background] Margolius D, Wong J, Goldman ML, Rouse-Iniguez J, Bodenheimer T. Delegating responsibility from clinicians to nonprofessional personnel: the example of hypertension control. J Am Board Fam Med. 2012 Mar-Apr;25(2):209-15. doi: 10.3122/jabfm.2012.02.100279. PMID 22403202